CLINICAL TRIAL: NCT05222269
Title: A Prospective, International, Multi-centre, Open-label, Single-arm Phase II Study Investigating the Predictive Value of [68Ga]Ga PentixaFor PET Imaging in Primary and Isolated Secondary CNS Lymphoma Patients
Brief Title: [68Ga]Ga-PentixaFor PET Imaging in CNS Lymphoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was early terminated due to low patient recruitment in already activated sites and difficult approval process in some of the anticipated countries. Thus, recruitment of the planned patient numbers in a reasonable time cannot be expected.
Sponsor: Pentixapharm AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTF202
Record Dates: First submitted 2022-01-05; First posted 2022-02-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2023-05

CONDITIONS: CNS Lymphoma
MeSH Terms: interventions — 68Ga-pentixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-PTF (Experimental): 150 (+/-50) Megabecquerel (MBq) 68Ga-PTF will be injected intravenously at three timepoints during the course of the standard of care treatment.
  Interventions: Drug: 68Ga-PTF

INTERVENTIONS:
Drug: 68Ga-PTF — 68Ga-PTF will be injected intravenously at three time points during the course of the standard treatment of the patient.
  Other Names: 68Ga-PentixaFor

SUMMARY:
This will be an open, single-arm, international, multicentre, phase II imaging study to assess the predictive value of [68Ga]Ga PentixaFor PET imaging in primary and isolated secondary central nervous system lymphoma (CNSL) patients scheduled to undergo induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained according to international guidelines and local laws by patient (or legally acceptable representative, if the patient is temporarily legally not competent owing to his/her disease). [Note: No invasive study-specific procedures may be carried out until this consent has been given.]
2. Patient aged 18 years or above (either sex).
3. Histologically confirmed primary or secondary CNSL based on cytology/flow cytometry of cerebrospinal fluid (CSF) or brain biopsy.
4. Disease exclusively located in the CNS (primary CNSL or secondary CNSL with isolated CNS relapse). Subjects who had undergone allogeneic stem cell transplant > 12 months prior to first dose of study drug, have no evidence of active graft versus host disease, and are not on systemic immunosuppressive therapy are allowed to participate in the study.
5. At least one measurable parenchymal lesion. [Note: parenchymal CNSL is a "must", and additional locations such as leptomeningeal disease are permitted.]
6. Previously untreated CNS disease. [Note: Previous or ongoing steroid treatment is permitted. Prophylaxis chemotherapy is not necessary, as induction chemotherapy will start within 72 hours after PTF-PET.]
7. At least one morphologically measurable lesion according to the IPCG criteria (Appendix 1).
8. Patients scheduled to undergo induction chemotherapy based on one of the following:

   High-dose methotrexate (HD-MTX)-based chemotherapy, ICE/DeVIC or High-dose cytarabine (HD-AraC)-based chemotherapy.
9. ECOG performance status ≤ 2 for patients aged ≥65 years; ECOG performance status ≤ 3 for patients aged <65 years.
10. Life expectancy of at least 3 months, as estimated by the investigator.
11. For women of child-bearing potential: negative pregnancy test.
12. For sexually active female patients of child-bearing potential: The patient agrees to take adequate contraceptive measures during study participation and also agrees to continue use of this method for the duration of the study and for 6 months after the last dose of PTF.
13. For male patients whose partner is of child-bearing potential: The patient is willing to ensure that he and his partner use effective contraception during the study and for 6 months after the last dose of PTF.

Exclusion Criteria:

1. Known hypersensitivity to [68Ga]Ga-PentixaFor or its components.
2. Contraindication for contrast-enhanced MRI as set out in the relevant institutional guidelines (e.g., pacemaker, defibrillator, aneurysm clip, metal in the body, renal insufficiency, severe claustrophobia etc.).
3. Contraindication for the use of gadolinium contrast for MRI.
4. Contraindication for PET according to institutional guidelines (weight-based, e.g. weight > 180 kg).
5. Inability to lie still for the entire imaging time.
6. Systemic lymphoma manifestation (outside the CNS).
7. Presence of active infection at screening or history of serious infection within the previous 6 weeks (except HIV infection: patients with HIV-associated primary CNSL are considered eligible).
8. Administration of another investigational medicinal product within the 30 days (or 5 excretion half-lives, whichever period is the longer) before first treatment with PTF.

   [Note: Re screening may be performed to accept washout of prior agents.]
9. Current toxicity of Grade >2 from previous standard or investigational therapies (grade according to the NCI Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0).
10. For female patients: Pregnancy (existing or intended) or breast-feeding.
11. Renal impairment: Both of the following:

    Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2 Creatinine clearance < 60 ml/min
12. Hepatic impairment: Both of the following:

    Aspartate aminotransferase (AST) > 3x upper limit of normal Alanine aminotransferase (ALT) > 3x upper limit of normal
13. Presence of any unstable systemic disease (including, but not limited to, active infection, uncontrolled hypertension, unstable angina, congestive heart failure, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease.
14. Presence of psychiatric disease, alcohol abuse or any other medical condition(s) that, in the opinion of the investigator, makes the patient unable to comply with study procedures and visits.
15. Patient weight ≤ 48 kg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of interim 68Ga-PTF-PET (after 6 ± 2 weeks of induction chemotherapy) for progression-free survival (PFS) | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  68Ga-PTF PET negativity for CXCR4 will be determined by visual analysis in central reading. For PFS assessment (yes/no variable), tumour progression or relapse will be determined according to the IPCG response criteria (Abrey et al. 2005) for the time period starting at baseline and ending at approx. 12 months after induction chemotherapy completion.
  The negative predictive value is defined as follows: Number of patients without tumour progression or relapse / number of patients with interim 68Ga-PTF PET assessed as CXCR4-negative by central reviewer. The proportion obtained will be multiplied by 100 to obtain a percentage value.
  This NPV will be calculated for the entire study population and also stratified by induction chemotherapy regimen (HD-MTX-based, DeVIC/ICE, HD-AraC-based regimen).

SECONDARY OUTCOMES:
Positive predictive value (PPV) of interim 68Ga-PTF PET (after 6 ± 2 weeks of induction chemotherapy) for PFS | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  68Ga-PTF PET positivity for CXCR4 will be determined by visual analysis in central reading. For PFS assessment (yes/no variable), tumour progression or relapse will be determined according to the IPCG response criteria (Abrey et al. 2005) for the time period starting at baseline and ending at approx. 12 months after induction chemotherapy completion.
  The positive predictive value is defined as follows: Number of patients with tumour progression or relapse / number of patients with interim 68Ga-PTF PET assessed as CXCR4-positive by central reviewer. The proportion obtained will be multiplied by 100 to obtain a percentage value.
Frequency and severity of AEs | up to 6 months
  The safety will be reported by frequency, system organ class categories, and severity of adverse events (AEs). The numbers and proportions of patients with any treatment-emergent adverse event (TEAE), and any serious TEAE will be summarized.
Predictive values of 68Ga-PTF PET at the end of induction chemotherapy for PFS | end of induction chemotherapy up to 12 months after induction chemotherapy completion
  The negative predictive value (NPV) and the positive predictive value (PPV) for the prediction of PFS at the end of induction chemotherapy will be determined as described in outcome 1 and 2.
Predictive values of 68Ga-PTF PET at interim examination (after 6 ± 2 weeks of induction chemotherapy) and end-of-chemotherapy-treatment for complete response (CR) | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  NPV of interim (after 6 ± 2 weeks of induction chemotherapy) 68Ga-PTF PET for the prediction of 16(±1) months CR.
  PPV of interim (after 6 ± 2 weeks of induction chemotherapy) 68Ga-PTF PET for the prediction of 16(±1) months CR.
  NPV of end-of-chemotherapy 68Ga-PTF PET for the prediction of 16(±1)-months CR.
  PPV of end-of-chemotherapy 68Ga-PTF PET for the prediction of 16(±1)-months CR.
  Response assessment will be performed 12 months after completion of induction chemotherapy and predictive values will be calculated with the results from the central visual analysis of the 68Ga-PTF PET scans at the different timepoints of induction chemotherapy.
Maximum standardized uptake value (SUVmax), SUVpeak and SUV mean | after pretreatment examination up to 12 months after induction chemotherapy completion (end of follow-up period)
  Maximum standardized uptake value (SUVmax), SUVpeak and SUV mean will be determined for the pre-treatment 68Ga-PTF scan and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Maximum tumour-to background ratio (TBRmax) and TBRmean | after pretreatment examination up to 12 months after induction chemotherapy completion (end of follow-up period)
  Maximum tumour-to background ratio (TBRmax) and TBRmean will be determined for the pre-treatment 68Ga-PTF scan and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Metabolic tumour volume (MTV) | after pretreatment examination up to 12 months after induction chemotherapy completion (end of follow-up period)
  Metabolic tumour volume (MTV) will be determined for the pre-treatment 68Ga-PTF scan by relative and fixed thresholding method and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Maximum standardized uptake value (SUVmax), SUVpeak and SUV mean | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  Maximum standardized uptake value (SUVmax), SUVpeak and SUV mean will be determined for the interim 68Ga-PTF scan and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Maximum tumour-to background ratio (TBRmax) and TBRmean | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  Maximum tumour-to background ratio (TBRmax) and TBRmean will be determined for the interim 68Ga-PTF scan and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Metabolic tumour volume (MTV) | after 6 +/-2 weeks of induction chemotherapy (interim examination) up to 12 months after induction chemotherapy completion (end of follow-up period)
  Metabolic tumour volume (MTV) will be determined for the interim 68Ga-PTF scan by relative and fixed thresholding method and will be analyzed for their association with 16(±1)-months PFS and also with 16(±1) months CR.
Predictive values of changes between pre-treatment and interim 68Ga-PTF PET imaging parameters for PFS | From visit 2 (first 68Ga-PTF PET) up to 12 months after induction chemotherapy completion
  The association of ΔSUVmax (change in SUVmax between pre-treatment 68Ga-PTF PET and interim 68Ga PTF PET) with 16(±1)-months PFS will be determined
Sensitivity of pre-treatment 68Ga-PTF PET for CXCR4-positivity | up to 12 months after induction chemotherapy completion
  In the fraction of patients from whom biopsy tissue is available, the sensitivity of the pre-treatment 68Ga-PTF PET to detect CXCR4 overexpression by immunohistochemistry (IHC) will be determined centrally on a patient basis
Concordance in the classification as CNSL-suspect ('yes'/'no') by 68Ga-PTF PET and MRI at baseline, on a patient level | after Visit 4 (after 6 +/-2 weeks of induction chemotherapy)
  Diagnostic agreement between 68Ga-PTF PET and MRI at baseline imaging (after 6 +/-2 weeks of induction chemotherapy) will be determined on a patient level by evaluation of the concordance in the classification as CNSL-suspect ('yes'/'no') by 68Ga-PTF PET and MRI at baseline.
Comparison of lesion numbers categorised as CNSL-suspect by 68Ga-PTF PET and MRI at baseline | after Visit 4 (after 6 +/-2 weeks of induction chemotherapy)
  Diagnostic agreement between 68Ga-PTF PET and MRI at baseline imaging (after 6 +/-2 weeks of induction chemotherapy) will be determined on a patient level by comparing lesion numbers categorised as CNSL-suspect by 68Ga-PTF PET and MRI at baseline
Observer agreement of 68Ga-PTF PET (inter- and intra-reader agreement) | through study completion, an average of 6 months
  The following will be calculated with respect to 68Ga-PTF-PET positivity:
  1. Inter-reader agreement for pre-treatment 68Ga-PTF PET
  2. Inter-reader agreement for interim 68Ga-PTF PET
  3. Inter-reader agreement for 68Ga-PTF PET after induction chemotherapy completion
  4. Intra-reader agreement for pre-treatment 68Ga-PTF PET
  5. Intra-reader agreement for interim 68Ga-PTF PET
  6. Intra-reader agreement for 68Ga-PTF PET after induction chemotherapy completion
  7. Overall inter-reader agreement
  8. Overall intra-reader agreement. The intra-reader assessment will be based on an appropriately sized sample of readings.

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Aalborg, Aalborg, Denmark
- University Hospital CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No